CLINICAL TRIAL: NCT02131350
Title: Combination Treatment of Intravitreal Ranibizumab, Focal/Grid Laser and Panretinal Photocoagulation in Patients With Diabetic Macula Edema
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Takao Hirano, Department of Ophthalmology Shinshu University School of Medicine, Shinshu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2617
Record Dates: First submitted 2014-04-22; First posted 2014-05-06 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Macula Edema
MeSH Terms: interventions — Light Coagulation; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ranibizumab with Photocoagulation (Experimental)
  Interventions: Procedure: Photocoagulation; Drug: Ranibizumab

INTERVENTIONS:
Procedure: Photocoagulation — Photocoagulation include focal/grid laser and/or panretinal photocoagulation
Drug: Ranibizumab

SUMMARY:
The purpose of this study is to evaluate the mean gain in best corrected visual acuity and the number of intravitreal ranibizumab (IVR) injections under the combination treatment of IVR, focal/grid laser and panretinal photocoagulation. Our hypothesis is that suitable photocoagulation decreases the number of IVR injections.

ELIGIBILITY:
Inclusion Criteria:

* stable medication for the management of diabetes within 3 months
* visual impairment due to focal or diffuse diabetic macula edema
* decreased vision due to diabetic macula edema and not other causes

Exclusion Criteria:

* concomitant conditions in the study eye that could prevent the improvement in VA on the study
* active intraocular inflammation or infection in either eye
* uncontrolled glaucoma in either eye
* treatment with antiangiogenic drugs in the study eye within 3 months
* history of stroke and uncontrolled hypertension

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
best corrected visual acuity | every month, up to 36 months
  Best corrected visual acuity is measured with Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity chart and analysed.

CONTACTS AND LOCATIONS:
Locations (1):
- Department ou Ophthalmology Shinshu University School of Medicine, Matsumoto, Nagano, Japan